CLINICAL TRIAL: NCT04340076
Title: Dose Reduction of the New Generation Biologicals (IL17 and IL23 Inhibitors) in Psoriasis: A Pragmatic, Multicentre, Randomized, Controlled, Non-inferiority Study - BeNeBio Study
Brief Title: Dose Reduction of IL17 and IL23 Inhibitors in Psoriasis
Acronym: BeNeBio
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Belgium Health Care Knowledge Centre (Other Government); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80-85200-98-18562; 2019-004230-42 (EudraCT Number)
Record Dates: First submitted 2020-03-20; First posted 2020-04-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis; Psoriasis Vulgaris
Keywords: skin diseases; skin diseases (papulosquamous); biologicals; IL17 inhibitors; IL23 inhibitors; dose reduction
MeSH Terms: conditions — Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous | interventions — secukinumab; ixekizumab; brodalumab; guselkumab; risankizumab; tildrakizumab; bimekizumab

STUDY DESIGN:
Intervention Model Description: A multicentre, pragmatic, randomized, controlled, non-inferiority trial. Patients will be randomized 2:1 to dose reduction and usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose reduction (Experimental): Dose reduction by interval prolongation in 2 steps to a maximum decrease of 50% of the original dose when disease activity (PASI) and quality of life index (DLQI) remain low.
  Interventions: Drug: Secukinumab; Drug: Ixekizumab; Drug: Brodalumab; Drug: Guselkumab; Drug: Risankizumab; Drug: Tildrakizumab; Drug: Bimekizumab
- Normal dose (Active Comparator): Patients will continue treatment with the normal/maintenance dose of the biologicals.
  Interventions: Drug: Secukinumab; Drug: Ixekizumab; Drug: Brodalumab; Drug: Guselkumab; Drug: Risankizumab; Drug: Tildrakizumab; Drug: Bimekizumab

INTERVENTIONS:
Drug: Secukinumab — Maintenance/normal dose is 300 mg/4 weeks. First dose reduction step: 300 mg/6 weeks. Second dose reduction step: 300 mg/8 weeks.
  Other Names: Cosentyx
Drug: Ixekizumab — Maintenance/normal dose is 80 mg/4 weeks. First dose reduction step: 80 mg/6 weeks. Second dose reduction step: 80 mg/8 weeks
  Other Names: Taltz
Drug: Brodalumab — Maintenance/normal dose is 210 mg/2 weeks. First dose reduction step: 210 mg/3 weeks. Second dose reduction step: 210 mg/4 weeks.
  Other Names: Kyntheum
Drug: Guselkumab — Maintenance/normal dose is 100 mg/8 weeks. First dose reduction step: 100 mg/12 weeks. Second dose reduction step: 100 mg/16 weeks.
  Other Names: Tremfya
Drug: Risankizumab — Maintenance/normal dose is 150 mg every 12 weeks. First dose reduction step: 150mg/18 weeks. Second dose reduction step: 150mg/24 weeks.
  Other Names: Skyrizi
Drug: Tildrakizumab — Maintenance/normal dose is 100 mg or 200 mg every 12 weeks. First dose reduction step: 100 mg or 200 mg/18 weeks. Second dose reduction step: 100 mg or 200 mg/24 weeks.
  Other Names: Ilumetri
Drug: Bimekizumab — Maintenance/normal dose is 320 mg/8 weeks. First dose reduction step: 320 mg/12 weeks. Second dose reduction step: 320 mg/16 weeks.
  Other Names: Bimzelx

SUMMARY:
The main objective of this study is to investigate whether controlled dose reduction of IL17 or IL23 inhibiting biologics is not inferior compared to usual care in psoriasis patients. Therefore, a pragmatic, multicentre, randomized, controlled, non-inferiority study will be carried out.

DETAILED DESCRIPTION:
Rationale: Biologics are very effective treatments for psoriasis. Research indicated that the dose of TNFα-blocking biologics can be reduced in a proportion of patients. Safety profiles can improve and costs can be reduced if the reduction of the dose is successful. Recently, the newest generation of biologics entered the market: interleukin (IL) 17 and IL23 inhibitors. It is not yet known whether dose reduction of these agents is possible, and to what extent they can be reduced. The timely investigation of the possibilities for dose reduction of new biologics is therefore important.

Objectives: The primary goal is to investigate whether controlled dose reduction of IL17 or IL23 inhibiting biologics is not inferior compared to usual care. This is measured by comparing the proportion of long-term disease flares between the two groups (dose reduction group versus usual care group). Secondary goals are: determining the proportion of patients with successful dose reduction, clinical effectiveness measured with the Psoriasis Area and Severity score (PASI) score, Dermatology Life Quality Index (DLQI) scores, predictors for successful dose reduction, safety, and cost-effectiveness of dose reduction. Pharmacokinetic (PK) analysis will be performed for modeling.

Study design: a multicenter, practice-oriented, pragmatic, randomized, controlled, non-inferiority study.

Study population: Patients treated with the newest generation of biologics (IL17 or IL23 inhibitors), with long-term stable low disease activity at a normal dose. A total of 244 patients will be randomized (2:1) to dose reduction or continuation of usual care.

Intervention: Dose reduction by interval prolongation in 2 steps to a maximum decrease of 50% of the original dose when disease activity (PASI) and quality of life index (DLQI) remain low.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis (primarily)
* Treatment for at least 6 months with IL23 or IL17 inhibitor in a normal dose (dose advised by the label)
* PASI≤ 5 at inclusion and in previous 6 months (if no PASI scores are available, it should be clear from the patient record that psoriasis was clear/almost clear in previous 6 months).
* DLQI ≤ 5 at inclusion

Exclusion Criteria:

* Another indication than plaque psoriasis as the main indication for biologic use (e.g. patient receives biologic for rheumatoid arthritis as the main indication).
* Concomitant use of systemic immunosuppressants other than methotrexate or acitretin (e.g. prednisone, cyclosporine etc).
* Severe comorbidities with short life-expectancy (e.g. metastasized tumor).
* Presumed inability to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the incidence proportion of persistent flares (Psoriasis Area and Severity Index (PASI) >5 for ≥ 3 months). | 18 months

SECONDARY OUTCOMES:
Whether participants will have successful DR after 12 and 18 months, defined as using a lower dose than the normal dose and PASI ≤ 5. | 18 months
  Definition of successful dose reduction: lower dose than the normal dose and PASI≤ 5.
Psoriasis disease activity, measured with the Psoriasis Area and Severity Index (PASI) at each 3-monthly study visit. | 18 months
Dermatology-related quality of life as measured with the Dermatology Life Quality Index (DLQI) at each 3-montly study visit. | 18 months
Whether participants will have short disease flares throughout the study period (18 months), defined as a PASI > 5 at one time point. | 18 months
Whether other anti-psoriatic medication will be initiated in participants during the study period (18 months). | 18 months
Whether participants will have serious adverse events (SAE) and adverse events of special interest (AEoSI) during the study period. | 18 months
  AEoSI include, but are not limited to, infections, malignancies, and joint complaints or new-onset psoriatic arthritis.
Drug trough levels of each included drug, measured in blood serum samples which will be collected from participants at each 3-montly time point. | 18 months
Anti-drug antibody levels of each included drug, measured in blood serum samples which will be collected from participants at each 3-montly time point. | 18 months
Utilities, derived from EuroQoL 5 Dimensions (EQ-5D-5L) questionnaires, which will be measured at each 3-montly time point. | 18 months
  Utility scores will be used to calculate quality adjusted life years (QALYs) which are used to determine cost-effectiveness of DR.
Health status of participants, assessed by using the Short Form 36 (SF-36) version 2 questionnaire at every 3-monthly time point. | 18 months
Volumes of care, as measured with the iMTA Medical Consumption Questionnaire (MCQ) at each 3-monthly time point. Scores will be used to calculate direct medicals costs and non-medical costs. | 18 months
Loss of productivity and presenteeism of participants, as measured with the iMTA Productivity Cost Questionnaire (PCQ) at each 3-monthly time point. Scores will be used to calculate direct medicals costs and non-medical costs. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Elke de Jong, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (19):
- Belgium (8):
  - ULB Erasme, Brussels
  - Ghent University Hospital, Ghent
  - AZ Maria Middelares, Ghent
  - AZ St Lucas, Ghent
  - UCL Saint Luc, Leuven
  - UZ Leuven, Leuven
  - CHU Liege, Liège
  - Dermatologie Maldegem, Maldegem
- Netherlands (11):
  - Ziekenhuisgroep Twente, Almelo
  - Bravis hospital, Bergen op Zoom
  - Amphia Hospital, Breda
  - Slingeland hospital, Doetinchem
  - Catharina hospital, Eindhoven
  - UMC Groningen, Groningen
  - Maastricht UMC, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
  - Máxima Medisch Centrum, Veldhoven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Schoot LS, van den Reek JMPA, Grine L, Schots L, Kievit W, Lambert JLW, de Jong EMGJ. Dose reduction of the new generation biologics (IL-17 and IL-23 inhibitors) in psoriasis: study protocol for an international, pragmatic, multicenter, randomized, controlled, non-inferiority study-the BeNeBio study. Trials. 2021 Oct 16;22(1):707. doi: 10.1186/s13063-021-05681-z. PMID 34656148